CLINICAL TRIAL: NCT02621320
Title: Effect of Vitamin D3 Supplementation on Exercise Performance in Wheelchair Athletes.
Brief Title: Vitamin D Supplementation in Wheelchair Indoor Athletes
Acronym: VitD_SCI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Swiss Paraplegic Research, Nottwil (Network)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2015-11
Record Dates: First submitted 2015-11-24; First posted 2015-12-03 (Estimated); Last update posted 2016-11-22 (Estimated); Status verified 2016-11

CONDITIONS: Vitamin D Deficiency; Spinal Cord Injury; Drug Effects; Dietary Supplements; Physical Education and Training/Methods
Keywords: Vitamin D; Exercise Performance; Wheelchair Athletes; Indoor sports; Wingate; Isokinetic Dynamometer
MeSH Terms: conditions — Vitamin D Deficiency; Spinal Cord Injuries | interventions — Vitamin D

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vitamin D (Experimental): alcohol-based (Ethanol 65%) Vitamin D3 (Vi-De 3®. WILD) solution 6000IU per day.
  Interventions: Dietary Supplement: Vitamin D
- Placebo (Placebo Comparator): Same alcohol-based solution (Ethanol 65%) as intervention product but without cholecalciferol
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Vitamin D — Vitamin D3 (Vi-De 3®. WILD) 6000IU daily over a period of 12 weeks.
  Arms: Vitamin D
Dietary Supplement: Placebo — alcohol-based solution 1.3ml daily over a period of 12 weeks.
  Arms: Placebo

SUMMARY:
There is a high prevalence of vitamin D deficiency in Switzerland. In indoor-athletes as well as wheelchair users, vitamin D deficiency occurs even more often. It is well established that vitamin D deficiency has a negative effect on health. However, vitamin D supplementation in individuals with a vitamin D deficiency has a positive effect on muscle performance. In recently published studies with able-bodied subjects, it has been shown that a normal vitamin D level (>75nmol/L) can only be achieved with a high-dose supplementation of vitamin D.

The aim of this study is to examine the effect of vitamin D supplementation on exercise performance in wheelchair athletes with vitamin D deficiency . All participants with a vitamin D deficiency are assigned to the intervention group and treated with 6000 IU of vitamin D3 daily over a period of 12 weeks. All participants who have a normal vitamin D level will receive placebo treatment (control group). The physical performance is measured three times at baseline, after six weeks and 12 weeks. The measurements include a Wingate and a dynamometer test.

ELIGIBILITY:
Inclusion Criteria:

* swiss elite wheelchair athlete
* 18 to 60 years
* male, healthy
* at least 2x45min sports a week

Exclusion Criteria:

* participation in another study
* medication which influences performance
* respiratory and cardiovascular disease
* daily intake of >400IU Vitamin D
* parathyroid gland disease
* kidney insufficiency
* visit abroad below the 37th parallel latitude during study or shortly before

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2015-11; Primary Completion 2016-07 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
peak power | delta change from pre to 12 weeks post supplementation
  peak power measured during wingate test
maximum torque | delta change from pre to 12 weeks post supplementation
  maximum torque measured with dynamometer

SECONDARY OUTCOMES:
Vitamin D serum level | week 0, 1 day before they start supplementation
  measured with venous blood sample
Vitamin D serum level | 12 weeks post supplementation
  measured with venous blood sample
Count of injuries | 12 weeks post supplementation
  DASH questionaire

OTHER OUTCOMES:
Heart rate | week 0, 1 day before they start supplementation
  Peak heart rate measured during wingate test
Heart rate | 12 weeks post supplementation
  Peak heart rate measured during wingate test
blood lactate concentration | week 0, 1 day before they start supplementation
  before, during and after wingate test
blood lactate concentration | 12 weeks post supplementation
  before, during and after wingate test

CONTACTS AND LOCATIONS:
Locations (1):
- Swiss Paraplegic Centre, Nottwil, Canton of Lucerne, Switzerland